CLINICAL TRIAL: NCT04231214
Title: Acute and Two-week Effects of Spiolto® Respimat® (Tiotropium/Olodaterol) on Cardiac Function, the Autonomic Nervous System and Small Airway Function in Hyperinflated COPD Subjects
Brief Title: Effects of Spiolto® Respimat® (Tiotropium/Olodaterol) on Cardiac Function in Hyperinflated COPD Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 19-01 SPIOMI
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — tiotropium-olodaterol

STUDY DESIGN:
Intervention Model Description: Spiolto® Respimat® or nebulized 0.9 % saline on Day 1 and Day 9, followed by two weeks open label self-administration of Spiolto® Respimat®
Who Masked: Investigator, Outcomes Assessor
Masking Description: Staff at study site and data analysts are blinded for the primary endpoint (acute effects of Spiolto® Respimat® on cardiac function)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment sequence 1 (Experimental): Spiolto® Respimat® on Day 1 0.9% nebulized saline on Day 9 Spiolto® Respimat® from Day 10 to Day 24
  Interventions: Drug: Olodaterol-Tiotropium
- Treatment sequence 2 (Experimental): 0.9% nebulized saline on Day 1 Spiolto® Respimat® on Day 9 Spiolto® Respimat® from Day 10 to Day 24
  Interventions: Drug: Olodaterol-Tiotropium

INTERVENTIONS:
Drug: Olodaterol-Tiotropium — 5µg Olodaterol and 5 µg Tiotropium via the soft mist inhaler Respimat®, administered once on Day 1 or Day 9 and daily from Day 10 to Day 24

SUMMARY:
The purpose of this study is to examine the effect of a combined LABA/LAMA treatment with olodaterol/tiotropium on small airway function, autonomic nervous system and cardiac function in COPD. The main objective is to study the acute effect of dual bronchodilation with olodaterol/tiotropium on cardiac function measured by MRI. This work is unique as it assesses the effects of Spiolto® Respimat® on the left-ventricular end-diastolic volume and muscle sympathetic nerve activity, two endpoints relevant for cardiovascular disease. Furthermore, the study concept introduces exhaled particle analysis as a measure for small airway function, thus offering the opportunity for a mechanistic link between airway openness, hyperinflation, and cardiac function.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to give written informed consent.
* Male and female subjects, aged ≥ 40 years. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart), and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is post-menopausal, with documented proof of hysterectomy or tubal ligation, or meets clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after treatment -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
* Subjects with stable COPD according to the current GOLD guidelines (GOLD 2018).
* Subjects with airflow limitation indicated by a post-bronchodilator FEV1 <80% of the predicted normal value and a post-bronchodilator FEV1/FC<0.7 at Visit 1. Post-bronchodilator refers to within 10-15 min after inhalation of 400 µg (4x100 µg) of salbutamol.
* Current or ex-smokers who have a smoking history of at least 10 pack years. (Ten pack-years are defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.)
* Hyperinflated subjects with RVol>135% predicted as measured at Visit 1, before intake of salbutamol.

Exclusion Criteria:

* Any clinically relevant abnormal findings in physical examination, clinical chemistry, haematology, urinalysis, vital signs, lung function or ECG at screening visit, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study or may influence the results of the study, or the subject's ability to participate in the study.
* Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease (including but not confined to aneurysm, hypokalemia, decompensated heart failure or hypertrophic obstructive cardiomyopathy), malignancy, hepatic disease, renal disease, haematological disease, neurological disease, endocrine disease (including but not confined to thyrotoxicosis) or pulmonary disease other than COPD (including but not confined to tuberculosis, bronchiectasis, cystic fibrosis, pulmonary hypertension, sarcoidosis, interstitial lung disease or lung fibrosis).
* Use of other investigational drug (approved or unapproved) at the time of enrolment, or within 30 days or 5 half-lives prior to Visit 1, whichever is longer.
* History of drug or alcohol abuse.
* Risk of non-compliance with study procedures.
* Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study.
* History of an acute respiratory infection four weeks prior to Visit 1 and between Visit 1 and 3. These patients will not be eligible, but will be permitted to rescreened 4 weeks after the resolution of the respiratory tract infection.
* Subjects with conditions contraindicated for treatment with, or having a history of reactions/hypersensitivity to any of the following inhaled drugs, drugs of a similar class or any component thereof:

  * anticholinergics
  * long and short acting beta-2 agonists
  * sympathomimetic amines
* Subjects with a history of long QT syndrome or whose QTcF (Fridericia method) measured at Visit 1 is prolonged (>450 ms for males and >470 ms for females). These subjects should not be re-screened.
* Subjects who have clinically significant cardiovascular abnormalities, which could interfere with the assessment of the study treatment (such as but not limited to cardiac arrhythmias, heart failure with left ventricular ejection fraction < 40 % as determined by MRI scan at Visit 2, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, history of myocardial infarction 6 months prior to Visit 1 or uncontrolled hypertension)
* Subjects with a known history or current atrial fibrillation to be confirmed by ECG at Visit 1.
* Subjects with pacemaker or bypass.
* Subjects with extensive tattoos.
* Subjects with a mean sitting systolic blood pressure >160 mmHg and/or mean sitting diastolic blood pressure > 90 mmHg at Visit 1. These subjects will be permitted to be re-screened after initiation or intensification of an antihypertensive therapy and achieving a controlled disease status.
* History of malignancy of any organ system (other than localized basal cell carcinoma of the skin), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
* Subjects with narrow-angle glaucoma, symptomatic benign prostatic hyperplasia or bladder-neck obstruction or severe renal impairment (GFR ≤ 50 mL/min/1.73 m2) including those with end-stage renal disease requiring dialysis or urinary retention. Benign Prostatic Hyperplasia (BPH) subjects who are stable on treatment can be considered.
* Subjects with insulin-dependent diabetes mellitus.
* Clinically evident polyneuropathy.
* Subjects with active/ clinical history of asthma.
* Subjects unable to undergo MRI scans, including claustrophobia or presence of any metal objects within the patient, preventing from MRI scan (e.g. pacemaker, aneurysm clips).
* History of one COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization within 3 months prior to Visit 1, to 3. Subjects may be re-screened after a minimum of 3 months after the resolution of the COPD exacerbation.
* More than one COPD exacerbation that required treatment with antibiotics, systemic steroids (oral or intravenous) or hospitalization within one year before Visit 1.
* Subjects requiring long term oxygen therapy on a daily basis for chronic hypoxemia.
* Subjects with pulmonary lobectomy or lung volume reduction surgery or lung transplantation.
* Subjects with a pre-existing diagnosis of alpha-1 antitrypsin deficiency or an alpha-1 antitrypsin blood level below the normal range on Visit 1.
* Subjects with a body mass index (BMI) of more than 35 kg/m2.
* Subjects participating in or planning to participate in the active phase of a supervised pulmonary rehabilitation program during the study.
* Subjects receiving any medications in the classes listed in Table 8-1 and Table 8-2.
* Subjects receiving medications in the classes listed in Table 8-3 should be excluded unless the medication has been stable for the specified period and the stated conditions have been met.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

PRIMARY OUTCOMES:
Change from baseline in left ventricular enddiastolic volume index (LVEDVi) after single dose of Spiolto® Respimat® versus nebulized saline | Day -8 (baseline), Day 1, Day 9, Day 24
  Left ventricular enddiastolic volume index (LVEDVi) is a measurement of the volume of blood in the heart's left ventricular chamber at the end of the chamber's filling with blood and will be determined as measured by MRI

SECONDARY OUTCOMES:
Channge from baseline in left ventricular enddiastolic volume index (LVEDVi) multiple doses of Spiolto® Respimat® versus nebulized saline | Day 24
  Left ventricular enddiastolic volume index (LVEDVi) is a measurement of the volume of blood in the heart's left ventricular chamber at the end of the chamber's filling with blood and will be determined as measured by MRI. LVEDVi after multiple doses will be compared with LVEDVi after single dose and baseline.
Muscle sympathetic nerve activity (MSNA) evaluated by microneurography as bursts/ 100 heart beats after single dose administration of Spiolto® Respimat® versus nebulized saline | Day 1, Day 9
  Muscle sympathetic nerve activity (MSNA) is a measurement of the sympathetic tone and will be recorded from the peroneal nerve
Forced Expiratory Volume in one second expressed as percent of Vital Capacity [FEV1/VC%] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  FEV1/VC% will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Mid Forced Expiratory Flow 25/75 [MFEF 25/75, L/s] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  MFEF 25/75 will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Peak Expiratory Flow 50 [PEF, L/s] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  ´PEF will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Forced Expiratory Flow 50 [FEF 50, L/s] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  FEF 50 will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Forced Expiratory Flow 25 [FEF 25, L/s] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  FEF 25 will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Residual volume expressed as percent of Total Lung Capacity [RV/TLC%] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  RV/TLC% will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Forced Vital Capacity [FVC, volume] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  FVC will be measured by spirometry according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Inspiratory Capacity [IC, volume] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  IC will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Total Lung Capacity [TLC, volume] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  TLC will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Specific Airway Resistance [sRaw, kPa*s] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  sRaw will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Functional Residual Capacity [FRC, volume] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  FRC will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Slow Vital Capacity [SVC, volume] at baseline, after single dose and multiple of Spiolto® Respimat® versus nebulized saline. | Day -28, Day -8, Day 1, Day 9, Day 24
  SVC will be measured by bodyplethysmography according to the recommendations of the American Thoracic Society and the European Respiratory Society from 2005
Exhaled particle numbers per volume at baseline, after single dose and multiple dose of Spiolto® Respimat® versus nebulized saline. | Day -8, Day 1, Day 9, Day 24
  Exhaled particles will be collected using the particle collector device PExA by PExA AB, Göteborg, Sweden. A single breath aerosol analysis will be performed with a LASAIR particle counter.

CONTACTS AND LOCATIONS:
Locations (1):
- Fraunhofer ITEM, Hanover, Lower Saxony, Germany

IPD SHARING:
Plan to Share IPD: No